CLINICAL TRIAL: NCT03817008
Title: Impact of Ascending Aorta Replacement by Graft on Elastic Properties of Descending Thoracic Aorta Evaluated by Cardiac Magnetic Resonance Imaging
Brief Title: Changes in Elastic Properties of Descending Thoracic Aorta After Ascending Aorta Replacement
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier La Chartreuse (Other)
Collaborators: JAZAYERI Aline (Unknown); BOUCHOT Olivier (Unknown); JAZAYERI Saed (Unknown); MALAPERT Ghislain (Unknown); PETROSYAN Andreanik (Unknown)
Responsible Party: Principal Investigator, MORGANT Marie-Catherine, PI, Centre Hospitalier La Chartreuse
Other Study IDs: MORGANT 2019
Record Dates: First submitted 2019-01-17; First posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Aortic Surgery
MeSH Terms: interventions — Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Ascending aorta replacement with graft — Patient with planned Ascending aorta replacement with graft
  Other Names: cardiac MRI

SUMMARY:
The aim of our study was to evaluate the impact of aortic root replacement by a graft on the elastic properties of the descending thoracic aorta using cardiac Magnetic Resonance Imaging (MRI) and automatic post-processing.

Nineteen patients were operated on an aortic root aneurysm and a cardiac MRI allowing aortic compliance measurement was performed before and after surgery. Images were acquired with a 1.5 T MRI with only one additional sequence to a conventional aortic MRI protocol.

DETAILED DESCRIPTION:
Observational and retrospective trial on medical data only. The patients are operated of planned aortic root aneurysm without additional intervention.

The pre and postoperative cardiac MRI are planned in standard of care.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Elective patient
* Ascending aorta replacement with graft

Exclusion Criteria:

* Prior cardiac surgery
* Contraindication to performing cardiac MRI

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 19 patients operated in Cardiac Surgery unit of DIJON Hospital between September 2014 and December 2017.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
Aortic compliance of descending aorta (mm2/mmHg) | post-operative cardiac MRI performing between 12 and 24 months
  Aortic elastic properties of the descending aorta before and after aortic root replacement using cardiac MRI.
  Aortic compliance is a local measurement of elastic properties which is obtained with cardiac MRI images by computer processing.

SECONDARY OUTCOMES:
Aortic compliance of ascending aorta (mm2/mmHg) | post-operative cardiac MRI performing between 12 and 24 months
  Aortic elastic properties of the ascending aorta before and after aortic root replacement using cardiac MRI.
  Aortic compliance is a local measurement of elastic properties which is obtained with cardiac MRI images by computer processing.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morgant MC, Miteran J, Lin S, Laubriet A, Cochet A, Lalande A, Bouchot O. Impact of ascending aorta replacement by graft on elastic properties of descending thoracic aorta evaluated by cardiac magnetic resonance imaging. MAGMA. 2020 Oct;33(5):641-647. doi: 10.1007/s10334-020-00829-5. Epub 2020 Jan 31. PMID 32006121